CLINICAL TRIAL: NCT01072149
Title: A Three-way Incomplete Block Crossover Study to Investigate the 24-hour Pulmonary Function of Three Dosage Strengths of Fluticasone Furoate (FF)/GW642444 Inhalation Powder vs. Placebo, in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Study to Evaluate the Efficacy, Safety, Tolerability, Pharmacokinetic (PK), and Pharmacodynamic (PD) Profiles of 3 Doses of Fluticasone Furoate (FF)/GW642444 Inhalation Powder at the End of a 28-day Treatment Period in Subjects With Chronic Obstructive Pulmonary Disease (COPD) Compared to Placebo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 110946
Record Dates: First submitted 2010-02-12; First posted 2010-02-19 (Estimated); Results first posted 2013-12-25 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; Safety; FEV1; Efficacy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — fluticasone furoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 50mcg Fluticasone Furoate (FF)/25mcg GW642444 (Experimental): Inhaled Corticosteroid (ICS)/ Long Acting Beta Agonist(LABA)
  Interventions: Drug: Fluticasone Furoate (FF)/GW642444 Inhalation Powder
- 100mcg Fluticasone Furoate (FF)/25mcg GW642444 (Experimental): Inhaled Corticosteroid (ICS)/ Long Acting Beta Agonist(LABA)
  Interventions: Drug: Fluticasone Furoate (FF)/GW642444 Inhalation Powder
- 200mcg Fluticasone Furoate (FF)/25mcg GW642444 (Experimental): Inhaled Corticosteroid (ICS)/ Long Acting Beta Agonist(LABA)
  Interventions: Drug: Fluticasone Furoate (FF)/GW642444 Inhalation Powder
- placebo (Placebo Comparator): placebo
  Interventions: Device: placebo

INTERVENTIONS:
Drug: Fluticasone Furoate (FF)/GW642444 Inhalation Powder — Inhaled Corticosteroid (ICS)/ Long Acting Beta Agonist(LABA) for COPD
  Arms: 100mcg Fluticasone Furoate (FF)/25mcg GW642444; 200mcg Fluticasone Furoate (FF)/25mcg GW642444; 50mcg Fluticasone Furoate (FF)/25mcg GW642444
Device: placebo — placebo
  Arms: placebo

SUMMARY:
The Purpose of this study is to evaluate the 24-hour spirometry effect Forced Expiratory Volume in One second (FEV1) of 3 doses of Fluticasone Furoate (FF)/GW642444 Inhalation Powder at the end of a 28-day treatment period in subjects with Chronic Obstructive Pulmonary Disease (COPD) compared with placebo. Other objectives are to assess additional efficacy, plus the safety, pharmcodynamics and tolerability of concurrent treatment with Fluticasone Furoate (FF) plus GW642444 when administered at three dose levels for 28 days in subjects with COPD and to assess the steady-state pharmacokinetic profile of Fluticasone Furoatee (FF) and GW642444 at the end of each treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient/Inpatient; Male or female subjects
* Subjects must give their signed and dated written informed consent to participate.
* A female is eligible to enter and participate in the study if she is of: Non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is post-menopausal or surgically sterile). Surgically sterile females are defined as those with a documented hysterectomy and/or bilateral oophorectomy or tubal ligation. Post-menopausal females are defined as being amenorrhoeic, > 45 years, in the absence of hormone replacement therapy. However in questionable cases, a blood sample with FSH >40MIU/ml and estradiol < 40pg/ml (<140 pmol/L) is confirmatory.

OR

Child bearing potential, has a negative pregnancy test at screening, and agrees to one of the following acceptable contraceptive methods used consistently and correctly (i.e. in accordance with the approved product label and the instructions of the physician for the duration of the study - screening to follow-up contact):

* Complete abstinence from intercourse from screening until the follow-up contact; or
* Male partner is sterile (vasectomy with documentation of azoospermia) prior to female subject entry into the study, and this male partner is the sole partner for that subject; or
* Implants of levonorgestral inserted for at least 1 month prior to the study medication administration but not beyond the third successive year following insertion; or
* Injectable progestogen administered for at least 1 month prior to study medication administration; or
* Oral contraceptive (combined or progestogen only) administered for at least one monthly cycle prior to study medication administration; or
* Double barrier method: condom or occlusive cap (diaphragm or cervical/vault caps) plus spermicidal agent (foam/gel/film/cream/suppository); or
* An intrauterine device (IUD), inserted by a qualified physician, with published data showing that the highest expected failure rate is less than 1% per year; or
* Estrogenic vaginal ring; or
* Percutaneous contraceptive patches.
* Age: ≥40 years of age at Screening (Visit 1).
* COPD diagnosis: Subjects with a clinical history of COPD in accordance with the following definition by the American Thoracic Society/European Respiratory Society [Celli, 2004]: COPD is a preventable and treatable disease characterized by airflow limitation that is not fully reversible. The airflow limitation is usually progressive and is associated with an abnormal inflammatory response of the lungs to noxious particles or gases, primarily caused by cigarette smoking. Although COPD affects the lungs, it also produces significant systemic consequences.
* Tobacco use: subjects with a current or prior history of ≥10 pack-years of cigarette smoking at Screening (Visit 1). Former smokers are defined as those who have stopped smoking for at least 6 months prior to Screening (Visit 1).

Note: Pipe and/or cigar use cannot be used to calculate pack year history. Number of pack years = (number of cigarettes per day/20)) x number of years smoked

* Severity of Disease:
* Subject with a measured post-albuterol/salbutamol FEV1/FVC ratio of ≤0.70 at Screening (Visit 1). [Pelligrino, 2005]
* Subjects with a measured post-albuterol/salbutamol FEV1 ≤ 70% of predicted normal values calculated using NHANES III reference equations [Hankinson, 1999] at Screening (Visit 1). Post-bronchodilator spirometry will be performed approximately 10-15 minutes after the subject has self-administered 4 inhalations (i.e. total 400mcg.) of albuterol/salbutamol via an MDI with a valved-holding chamber. The FEV1/FVC ratio and FEV1 percent predicted values will be calculated by the centralized spirometry equipment.
* Dyspnea: Achieved a score of ≥2 on the Modified Medical Research Council Dyspnea Scale (mMRC, 0-4 scale) at Screening (Visit 1).

Exclusion Criteria:

* Pregnancy: Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* Asthma: Subjects with a current diagnosis of asthma. (Subjects with a prior history of asthma are eligible if they have a current diagnosis of COPD)
* α1-antitrypsin deficiency: Subjects with α-1 antitrypsin deficiency as the underlying cause of COPD
* Other respiratory disorders: Subjects with active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung diseases or other active pulmonary diseases
* Lung resection: Subjects with lung volume reduction surgery within the 12 months prior to Screening
* Chest X-ray (or CT scan): Subjects with a chest X-ray (or CT scan) thats reveals evidence of clinically significant abnormalities not believed to be due to the presence of COPD. A chest X-ray must be taken at Screening if a chest X-ray or CT scan is not available within 6 months prior to Screening (Visit 1)
* Hospitalization: Subjects who are hospitilized due to poorly controlled COPD with 12 weeks of Screening (Visit 1)
* Poorly controlled COPD: Subjects with poorly controlled COPD defined as the occurrence of any of the following in the 6 weeks prior to Screening (Visit 1):
* acute worsening of COPD that is managed by the subject with corticosteroids or antibiotics, or that requires treatment prescribed by a physician
* Lower respiratory tract infection: Subjects with lower respiratory tract infection that require the use of antibiotics within 6 weeks prior to Screening (Visit 1)
* Other diseases/abnormalities: Subjects with historical or current evidence of clinically significant cardiovascular (i.e., pacemaker), neurological, psychiatric, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or haematological abnormalities that are uncontrolled. Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
* Peptic Ulcer disease: Subjects with clinically significant peptic ulcer disease that is uncontrolled.
* Hypertension: Subjects with clinically significant hypertension that is uncontrolled
* Cancer: Subjects with carcinoma that has not been in complete remission for at least 5 years. Carcinoma in situ of the cervix, squamous cell carcinoma and basal cell carcinoma of the skin would not be excluded if the subject has been considered cured within 5 years since diagnosis.
* Drug/food allergy: Subjects with a history of hypersensitivity to any of the study medications (e.g. beta-agonists, corticosteroid) or components of the inhalation powder (e.g. lactose, magnesium stearate). In addition, patients with a history of severe milk protein allergy that, in the opinion of the study physician, contraindicates the subject's participation will also be excluded.
* Drug/alcohol abuse: Subjects with a known or suspected history of alcohol or drug abuse within the last 2 years
* Medication prior to spirometry: Subjects who are medically unable to withhold their albuterol/salbutamol or their ipratropium for the 4-hour period required prior to spirometry testing at each study visit.
* Additional medication: Use of certain medications such as bronchodilators and corticosteroids for the protocol-specific times prior to Visit 1 (the Investigator will discuss the specific medications)
* Oxygen therapy: Subjects receiving treatment with long-term oxygen therapy (LTOT) or nocturnal oxygen therapy required for greater than 12 hours a day. Oxygen prn use (i.e. ≤12 hours per day) is not exclusionary.
* Sleep apnea: Subjects with clinically significant sleep apnea who require use of continuous positive airway pressure (CPAP) device or non-invasive positive pressure ventilation (NIPPV) device.
* Pulmonary rehabilitation: Subjects who have participated in the acute phase of a
* Pulmonary Rehabilitation Program within 4 weeks prior to Screening or who will enter the acute phase of a Pulmonary Rehabilitation Program during the study. Subjects who are in the maintenance phase of a Pulmonary Rehabilitation Program are not excluded.
* Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures. Any infirmity, disability, or geographic location that would limit compliance for scheduled visits.
* Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study
* Prior use of study medication/other investigational drugs: Subjects who have previously been randomized in the Phase IIa (HZC111348 or B2C111045) study or Phase III (i.e. HZC112206, HZC112207, HZC102970, HZC102871) studies. Subjects who have received an investigational drug within 30 days of entry into this study (Screening), or within 5 drug half-lives of the investigational drug, whichever is longer
* Affiliation with investigator site: Study investigators, sub-investigators, study coordinators, employees of a participating investigator or immediate family members of the aforementioned are excluded from participating in this study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-01-01; Primary Completion 2010-07-01 (Actual); Study Completion 2010-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- United States (8):
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Madisonville, Kentucky
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Boscia JA, Pudi KK, Zvarich MT, Sanford L, Siederer SK, Crim C. Effect of once-daily fluticasone furoate/vilanterol on 24-hour pulmonary function in patients with chronic obstructive pulmonary disease: a randomized, three-way, incomplete block, crossover study. Clin Ther. 2012 Aug;34(8):1655-66.e5. doi: 10.1016/j.clinthera.2012.06.005. Epub 2012 Jul 11. PMID 22789766
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 110946 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110946 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110946 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110946 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110946 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 110946 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110946 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following screening and a 2-week Run-in Period, during which all participants received placebo, participants were randomized to receive 2 of the 3 strengths of study medication and placebo in the Treatment Phase of the study, which consisted of three 28-day treatment periods, each separated by a 14-day washout period.
Groups:
- Sequence 1: FF/VI 50/25 µg, Placebo, FF/VI 100/25 µg: Participants self-administered fluticasone furoate/vilanterol (FF/VI) 50/25 µg, placebo, and FF/VI 100/25 µg once every day (one inhalation in the morning) for 28 days via an Investigational Product Inhaler (IPI) during Treatment Periods 1, 2, and 3, respectively. The three treatment periods were separated by a 14-day washout period.
- Sequence 2: Placebo, FF/VI 100/25 µg, FF/VI 50/25 µg: Participants self-administered placebo, FF/VI 100/25 µg, and FF/VI 50/25 µg once every day (one inhalation in the morning) for 28 days via an IPI during Treatment Periods 1, 2, and 3, respectively. The three treatment periods were separated by a 14-day washout period.
- Sequence 3: FF/VI 200/25 µg, FF/VI 50/25 µg, Placebo: Participants self-administered FF/VI 200/25 µg, FF/VI 50/25 µg, and placebo once every day (one inhalation in the morning) for 28 days via an IPI during Treatment Periods 1, 2, and 3, respectively. The three treatment periods were separated by a 14-day washout period.
- Sequence 4: FF/VI 200/25 µg, Placebo, and FF/VI 100/25 µg: Participants self-administered FF/VI 200/25 µg, placebo, and FF/VI 100/25 µg once every day (one inhalation in the morning) for 28 days via an IPI during Treatment Periods 1, 2, and 3, respectively. The three treatment periods were separated by a 14-day washout period.
- Sequence 5: FF/VI 50/25 µg, FF/VI 100/25 µg, Placebo: Participants self-administered FF/VI 50/25 µg, FF/VI 100/25 µg, and placebo once every day (one inhalation in the morning) for 28 days via an IPI during Treatment Periods 1, 2, and 3, respectively. The three treatment periods were separated by a 14-day washout period.
- Sequence 6: FF/VI 50/25 µg, FF/VI 200/25 µg, Placebo: Participants self-administered FF/VI 50/25 µg, FF/VI 200/25 µg, and placebo once every day (one inhalation in the morning) for 28 days via an IPI during Treatment Periods 1, 2, and 3, respectively. The three treatment periods were separated by a 14-day washout period.
- Sequence 7: FF/VI 200/25 µg, Placebo, FF/VI 50/25 µg: Participants self-administered FF/VI 200/25 µg, placebo, and FF/VI 50/25 µg once every day (one inhalation in the morning) for 28 days via an IPI during Treatment Periods 1, 2, and 3, respectively. The three treatment periods were separated by a 14-day washout period.
- Sequence 8: Placebo, FF/VI 50/25 µg, FF/VI 100/25 µg: Participants self-administered placebo, FF/VI 50/25 µg, and FF/VI 100/25 µg once every day (one inhalation in the morning) for 28 days via an IPI during Treatment Periods 1, 2, and 3, respectively. The three treatment periods were separated by a 14-day washout period.
- Sequence 9: FF/VI 100/25 µg, FF/VI 50/25 µg, Placebo: Participants self-administered FF/VI 100/25 µg, FF/VI 50/25 µg, and placebo once every day (one inhalation in the morning) for 28 days via an IPI during Treatment Periods 1, 2, and 3, respectively. The three treatment periods were separated by a 14-day washout period.
- Sequence 10: FF/VI 100/25 µg, Placebo, FF/VI 50/25 µg: Participants self-administered FF/VI 100/25 µg, placebo, and FF/VI 50/25 µg once every day (one inhalation in the morning) for 28 days via an IPI during Treatment Periods 1, 2, and 3, respectively. The three treatment periods were separated by a 14-day washout period.
- Sequence 11: Placebo, FF/VI 200/25 µg, FF/VI 100/25 µg: Participants self-administered placebo, FF/VI 200/25 µg, and FF/VI 100/25 µg once every day (one inhalation in the morning) for 28 days via an IPI during Treatment Periods 1, 2, and 3, respectively. The three treatment periods were separated by a 14-day washout period.
- Sequence 12: Placebo, FF/VI 200/25 µg, FF/VI 50/25 µg: Participants self-administered placebo, FF/VI 200/25 µg, and FF/VI 50/25 µg once every day (one inhalation in the morning) for 28 days via an IPI during Treatment Periods 1, 2, and 3, respectively. The three treatment periods were separated by a 14-day washout period.
- Sequence 13: Placebo, FF/VI 100/25 µg, FF/VI 200/25 µg: Participants self-administered placebo, FF/VI 100/25 µg, and FF/VI 200/25 µg once every day (one inhalation in the morning) for 28 days via an IPI during Treatment Periods 1, 2, and 3, respectively. The three treatment periods were separated by a 14-day washout period.
- Sequence 14: FF/VI 200/25 µg, FF/VI 100/25 µg, Placebo: Participants self-administered FF/VI 200/25 µg, FF/VI 100/25 µg, and placebo once every day (one inhalation in the morning) for 28 days via an IPI during Treatment Periods 1, 2, and 3, respectively. The three treatment periods were separated by a 14-day washout period.
- Sequence 15: FF/VI 100/25 µg, FF/VI 200/25 µg, Placebo: Participants self-administered FF/VI 100/25 µg, FF/VI 200/25 µg, and placebo once every day (one inhalation in the morning) for 28 days via an IPI during Treatment Periods 1, 2, and 3, respectively. The three treatment periods were separated by a 14-day washout period.
- Sequence 16: Placebo, FF/VI 50/25 µg, FF/VI 200/25 µg: Participants self-administered placebo, FF/VI 50/25 µg, and FF/VI 200/25 µg once every day (one inhalation in the morning) for 28 days via an IPI during Treatment Periods 1, 2, and 3, respectively. The three treatment periods were separated by a 14-day washout period.
- Sequence 17: FF/VI 50/25 µg, Placebo, FF/VI 200/25 µg: Participants self-administered FF/VI 50/25 µg, placebo, and FF/VI 200/25 µg once every day (one inhalation in the morning) for 28 days via an IPI during Treatment Periods 1, 2, and 3, respectively. The three treatment periods were separated by a 14-day washout period.
- Sequence 18: FF/VI 100/25 µg, Placebo, FF/VI 200/25 µg: Participants self-administered FF/VI 100/25 µg, placebo, and FF/VI 200/25 µg once every day (one inhalation in the morning) for 28 days via an IPI during Treatment Periods 1, 2, and 3, respectively. The three treatment periods were separated by a 14-day washout period.
Period: Treatment Period 1 (28 Days)
Arm/Group | Sequence 1: FF/VI 50/25 µg, Placebo, FF/VI 100/25 µg | Sequence 2: Placebo, FF/VI 100/25 µg, FF/VI 50/25 µg | Sequence 3: FF/VI 200/25 µg, FF/VI 50/25 µg, Placebo | Sequence 4: FF/VI 200/25 µg, Placebo, and FF/VI 100/25 µg | Sequence 5: FF/VI 50/25 µg, FF/VI 100/25 µg, Placebo | Sequence 6: FF/VI 50/25 µg, FF/VI 200/25 µg, Placebo | Sequence 7: FF/VI 200/25 µg, Placebo, FF/VI 50/25 µg | Sequence 8: Placebo, FF/VI 50/25 µg, FF/VI 100/25 µg | Sequence 9: FF/VI 100/25 µg, FF/VI 50/25 µg, Placebo | Sequence 10: FF/VI 100/25 µg, Placebo, FF/VI 50/25 µg | Sequence 11: Placebo, FF/VI 200/25 µg, FF/VI 100/25 µg | Sequence 12: Placebo, FF/VI 200/25 µg, FF/VI 50/25 µg | Sequence 13: Placebo, FF/VI 100/25 µg, FF/VI 200/25 µg | Sequence 14: FF/VI 200/25 µg, FF/VI 100/25 µg, Placebo | Sequence 15: FF/VI 100/25 µg, FF/VI 200/25 µg, Placebo | Sequence 16: Placebo, FF/VI 50/25 µg, FF/VI 200/25 µg | Sequence 17: FF/VI 50/25 µg, Placebo, FF/VI 200/25 µg | Sequence 18: FF/VI 100/25 µg, Placebo, FF/VI 200/25 µg
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 2
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 1 (14 Days)
Arm/Group | Sequence 1: FF/VI 50/25 µg, Placebo, FF/VI 100/25 µg | Sequence 2: Placebo, FF/VI 100/25 µg, FF/VI 50/25 µg | Sequence 3: FF/VI 200/25 µg, FF/VI 50/25 µg, Placebo | Sequence 4: FF/VI 200/25 µg, Placebo, and FF/VI 100/25 µg | Sequence 5: FF/VI 50/25 µg, FF/VI 100/25 µg, Placebo | Sequence 6: FF/VI 50/25 µg, FF/VI 200/25 µg, Placebo | Sequence 7: FF/VI 200/25 µg, Placebo, FF/VI 50/25 µg | Sequence 8: Placebo, FF/VI 50/25 µg, FF/VI 100/25 µg | Sequence 9: FF/VI 100/25 µg, FF/VI 50/25 µg, Placebo | Sequence 10: FF/VI 100/25 µg, Placebo, FF/VI 50/25 µg | Sequence 11: Placebo, FF/VI 200/25 µg, FF/VI 100/25 µg | Sequence 12: Placebo, FF/VI 200/25 µg, FF/VI 50/25 µg | Sequence 13: Placebo, FF/VI 100/25 µg, FF/VI 200/25 µg | Sequence 14: FF/VI 200/25 µg, FF/VI 100/25 µg, Placebo | Sequence 15: FF/VI 100/25 µg, FF/VI 200/25 µg, Placebo | Sequence 16: Placebo, FF/VI 50/25 µg, FF/VI 200/25 µg | Sequence 17: FF/VI 50/25 µg, Placebo, FF/VI 200/25 µg | Sequence 18: FF/VI 100/25 µg, Placebo, FF/VI 200/25 µg
Started | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 2
Completed | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (28 Days)
Arm/Group | Sequence 1: FF/VI 50/25 µg, Placebo, FF/VI 100/25 µg | Sequence 2: Placebo, FF/VI 100/25 µg, FF/VI 50/25 µg | Sequence 3: FF/VI 200/25 µg, FF/VI 50/25 µg, Placebo | Sequence 4: FF/VI 200/25 µg, Placebo, and FF/VI 100/25 µg | Sequence 5: FF/VI 50/25 µg, FF/VI 100/25 µg, Placebo | Sequence 6: FF/VI 50/25 µg, FF/VI 200/25 µg, Placebo | Sequence 7: FF/VI 200/25 µg, Placebo, FF/VI 50/25 µg | Sequence 8: Placebo, FF/VI 50/25 µg, FF/VI 100/25 µg | Sequence 9: FF/VI 100/25 µg, FF/VI 50/25 µg, Placebo | Sequence 10: FF/VI 100/25 µg, Placebo, FF/VI 50/25 µg | Sequence 11: Placebo, FF/VI 200/25 µg, FF/VI 100/25 µg | Sequence 12: Placebo, FF/VI 200/25 µg, FF/VI 50/25 µg | Sequence 13: Placebo, FF/VI 100/25 µg, FF/VI 200/25 µg | Sequence 14: FF/VI 200/25 µg, FF/VI 100/25 µg, Placebo | Sequence 15: FF/VI 100/25 µg, FF/VI 200/25 µg, Placebo | Sequence 16: Placebo, FF/VI 50/25 µg, FF/VI 200/25 µg | Sequence 17: FF/VI 50/25 µg, Placebo, FF/VI 200/25 µg | Sequence 18: FF/VI 100/25 µg, Placebo, FF/VI 200/25 µg
Started | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 2
Completed | 3 | 2 | 1 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 2
Not Completed | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2 (14 Days)
Arm/Group | Sequence 1: FF/VI 50/25 µg, Placebo, FF/VI 100/25 µg | Sequence 2: Placebo, FF/VI 100/25 µg, FF/VI 50/25 µg | Sequence 3: FF/VI 200/25 µg, FF/VI 50/25 µg, Placebo | Sequence 4: FF/VI 200/25 µg, Placebo, and FF/VI 100/25 µg | Sequence 5: FF/VI 50/25 µg, FF/VI 100/25 µg, Placebo | Sequence 6: FF/VI 50/25 µg, FF/VI 200/25 µg, Placebo | Sequence 7: FF/VI 200/25 µg, Placebo, FF/VI 50/25 µg | Sequence 8: Placebo, FF/VI 50/25 µg, FF/VI 100/25 µg | Sequence 9: FF/VI 100/25 µg, FF/VI 50/25 µg, Placebo | Sequence 10: FF/VI 100/25 µg, Placebo, FF/VI 50/25 µg | Sequence 11: Placebo, FF/VI 200/25 µg, FF/VI 100/25 µg | Sequence 12: Placebo, FF/VI 200/25 µg, FF/VI 50/25 µg | Sequence 13: Placebo, FF/VI 100/25 µg, FF/VI 200/25 µg | Sequence 14: FF/VI 200/25 µg, FF/VI 100/25 µg, Placebo | Sequence 15: FF/VI 100/25 µg, FF/VI 200/25 µg, Placebo | Sequence 16: Placebo, FF/VI 50/25 µg, FF/VI 200/25 µg | Sequence 17: FF/VI 50/25 µg, Placebo, FF/VI 200/25 µg | Sequence 18: FF/VI 100/25 µg, Placebo, FF/VI 200/25 µg
Started | 3 | 2 | 1 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 2
Completed | 2 | 2 | 1 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 2 | 3 | 3 | 1 | 3 | 2
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3 (28 Days)
Arm/Group | Sequence 1: FF/VI 50/25 µg, Placebo, FF/VI 100/25 µg | Sequence 2: Placebo, FF/VI 100/25 µg, FF/VI 50/25 µg | Sequence 3: FF/VI 200/25 µg, FF/VI 50/25 µg, Placebo | Sequence 4: FF/VI 200/25 µg, Placebo, and FF/VI 100/25 µg | Sequence 5: FF/VI 50/25 µg, FF/VI 100/25 µg, Placebo | Sequence 6: FF/VI 50/25 µg, FF/VI 200/25 µg, Placebo | Sequence 7: FF/VI 200/25 µg, Placebo, FF/VI 50/25 µg | Sequence 8: Placebo, FF/VI 50/25 µg, FF/VI 100/25 µg | Sequence 9: FF/VI 100/25 µg, FF/VI 50/25 µg, Placebo | Sequence 10: FF/VI 100/25 µg, Placebo, FF/VI 50/25 µg | Sequence 11: Placebo, FF/VI 200/25 µg, FF/VI 100/25 µg | Sequence 12: Placebo, FF/VI 200/25 µg, FF/VI 50/25 µg | Sequence 13: Placebo, FF/VI 100/25 µg, FF/VI 200/25 µg | Sequence 14: FF/VI 200/25 µg, FF/VI 100/25 µg, Placebo | Sequence 15: FF/VI 100/25 µg, FF/VI 200/25 µg, Placebo | Sequence 16: Placebo, FF/VI 50/25 µg, FF/VI 200/25 µg | Sequence 17: FF/VI 50/25 µg, Placebo, FF/VI 200/25 µg | Sequence 18: FF/VI 100/25 µg, Placebo, FF/VI 200/25 µg
Started | 2 | 2 | 1 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 2 | 3 | 3 | 1 | 3 | 2
Completed | 2 | 2 | 0 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 2 | 2 | 3 | 1 | 3 | 2
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: All participants who self-administered placebo, FF/VI 50/25 µg, FF/VI 100/25 µg, or FF/VI 200/25 µg once every day (one inhalation in the morning) for 28 days via an IPI in any of the three 28-day treatment periods.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline data were collected in members of the Intent-to-Treat Population, comprised of all participants who had been randomized to and received at least one dose of randomised double-blind study medication in any treatment period.
  Years | 57.9 (9.24)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline data were collected in members of the Intent-to-Treat Population, comprised of all participants who had been randomized to and received at least one dose of randomised double-blind study medication in any treatment period.
  Participants
    Female | 29
    Male | 25
Race/Ethnicity, Customized [Number; unit: participants] — Baseline data were collected in members of the Intent-to-Treat Population, comprised of all participants who had been randomized to and received at least one dose of randomised double-blind study medication in any treatment period.
  participants
    African American/African Heritage | 6
    White | 48

OUTCOME MEASURES:

1. Primary Outcome: Time-adjusted Area Under the Curve (AUC) (i.e., Weighted Mean) for 24-hour Serial Forced Expiratory Volume in One Second (FEV1) at the End of Each 28-day Treatment Period
Description: FEV1 is defined as the amount of air that can be forcibly exhaled from the lungs in the first second of a forced exhalation. The weighted mean was calculated from pre-dose FEV1 (calculated as the mean of the -30 and -5 minute measurements) and post-dose FEV1 after 5, 15, 30, and 60 minutes and after 2, 4, 6, 8, 12, 16, 20, 22, 23, and 24 hours. Data are provided as the Least Squares Mean of the weighted mean for all three treatment periods. Analysis was performed using a mixed effects model with covariates of period treatment group, period Baseline, mean Baseline (defined as the mean of all available period Baseline FEV1 values), and period as fixed effects and participant as a random effect.
Time Frame: Pre-dose and the end of each 28-day treatment period (up to 19 weeks)
Population: Intent-to-Treat (ITT) Population: all participants who were randomized to and received at least one dose of trial medication in any treatment period. Only those participants available at the indicated time points were assessed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- Placebo: Participants self-administered placebo once every day (one inhalation in the morning) for 28 days via an Investigational Product Inhaler (IPI) during one of the three 28-day treatment periods.
- FF/VI 50/25 µg: Participants self-administered Fluticasone Furoate (FF) 50 micrograms (µg) and Vilanterol (VI) 25 µg as a dry powder once every day (one inhalation in the morning) for 28 days via an IPI during one of the three 28-day treatment periods.
- FF/VI 100/25 µg: Participants self-administered FF 100 µg and VI 25 µg as a dry powder once every day (one inhalation in the morning) for 28 days via an IPI during one of the three 28-day treatment periods.
- FF/VI 200/25 µg: Participants self-administered FF 200 µg and VI 25 µg as a dry powder once every day (one inhalation in the morning) for 28 days via an IPI during one of the three 28-day treatment periods.
Arm/Group | Placebo | FF/VI 50/25 µg | FF/VI 100/25 µg | FF/VI 200/25 µg
Number analyzed (Participants) | 48 | 32 | 30 | 30
Liters | 1.297 (0.0240) | 1.530 (0.0276) | 1.517 (0.0282) | 1.533 (0.0282)
Statistical Analysis 1: Comparison: Placebo vs FF/VI 50/25 µg; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Median Difference (Final Values) = 0.233, 95% CI 2-sided [0.179 to 0.287]
Statistical Analysis 2: Comparison: Placebo vs FF/VI 100/25 µg; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.220, 95% CI 2-sided [0.165 to 0.275]
Statistical Analysis 3: Comparison: Placebo vs FF/VI 200/25 µg; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.236, 95% CI 2-sided [0.181 to 0.291]

2. Secondary Outcome: Change From Period Baseline in Clinic Visit Trough FEV1 at the End of Each 28-day Treatment Period
Description: Trough FEV1 is defined as the mean of the 23- and 24-hour post-dose assessments. For each treatment period, period Baseline is defined as the mean of the -30 and -5 minute measurements taken on Period Day 1. Mean Baseline FEV1 for a given participant is defined as the mean of all available period Baseline FEV1 values. Data are presented as the mean of change from Baseline for all three treatment periods. Change from Baseline was calculated as the value at Period Day 29 minus the value at Baseline. Analysis was performed using a mixed effects model with covariates of period treatment group, period Baseline, mean Baseline, and period as fixed effects and participant as a random effect.
Time Frame: From Baseline to the end of each 28-day treatment period (up to 19 weeks)
Population: ITT Population. Only those participants available at the indicated time points were assessed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | FF/VI 50/25 µg | FF/VI 100/25 µg | FF/VI 200/25 µg
Number analyzed (Participants) | 48 | 32 | 30 | 30
Liters | -0.024 (0.0286) | 0.186 (0.0343) | 0.153 (0.0354) | 0.165 (0.0353)

3. Secondary Outcome: Change From Period Baseline in 25-hour Serial FEV1 at the End of Each 28 Day-treatment Period
Description: Change from period Baseline in 0-25 hour serial FEV1 (0 to 25 hours) over Period Days 28-29 was measured. Mean Baseline FEV1 for a given participant is defined as the mean of all available period Baseline FEV1 values. Data are presented as the mean of change from Baseline for all three treatment periods. Analysis was performed using a mixed effects repeated measures model with covariates of period treatment group, period Baseline, mean Baseline, period and time after dosing (nominal), in addition to time after dosing by period Baseline, time after dosing by mean Baseline, and time after dosing by period treatment interaction terms as fixed effects and participant as a random effect.
Time Frame: Baseline; pre-dose; 5 minutes, 15 minutes, 30 minutes, 60 minutes, and 2, 4, 6, 8, 12, 16, 20, 22, 23, 24, and 25 hours post-dose on Day 28 and Day 29 of each 28-day treatment period (up to 19 weeks)
Population: ITT Population. Only those participants available at the indicated time points were assessed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | FF/VI 50/25 µg | FF/VI 100/25 µg | FF/VI 200/25 µg
Number analyzed (Participants) | 49 | 32 | 31 | 31
Liters
  Mean pre-dose, n=49, 32, 31, 31 | -0.017 (0.0277) | 0.193 (0.0325) | 0.150 (0.0329) | 0.166 (0.0328)
  5 minutes, n=48, 32, 31, 31 | -0.002 (0.0289) | 0.208 (0.0340) | 0.186 (0.0344) | 0.217 (0.0343)
  15 minutes, n=46, 32, 31, 31 | 0.009 (0.0298) | 0.230 (0.0349) | 0.201 (0.0354) | 0.215 (0.0353)
  30 minutes, n=49, 32, 30, 31 | 0.006 (0.0304) | 0.255 (0.0359) | 0.200 (0.0365) | 0.240 (0.0363)
  60 minutes, n=49, 32, 30, 31 | -0.002 (0.0291) | 0.279 (0.0342) | 0.215 (0.0348) | 0.259 (0.0345)
  2 hours, n=49, 32, 30, 31 | -0.003 (0.0283) | 0.282 (0.0332) | 0.280 (0.0338) | 0.279 (0.0335)
  4 hours, n=49, 32, 30, 31 | -0.037 (0.0278) | 0.240 (0.0326) | 0.229 (0.0332) | 0.264 (0.0329)
  6 hours, n=49, 32, 30, 31 | -0.029 (0.0264) | 0.202 (0.0306) | 0.221 (0.0312) | 0.246 (0.0309)
  8 hours, n=49, 32, 30, 31 | -0.063 (0.0276) | 0.187 (0.0322) | 0.182 (0.0329) | 0.187 (0.0325)
  12 hours, n=48, 32, 30, 31 | -0.058 (0.0293) | 0.200 (0.0343) | 0.145 (0.0351) | 0.176 (0.0347)
  16 hours, n=48, 32, 29, 31 | -0.105 (0.0289) | 0.129 (0.0338) | 0.093 (0.0347) | 0.067 (0.0341)
  20 hours, n=48, 32, 30, 30 | -0.127 (0.0309) | 0.073 (0.0364) | 0.071 (0.0373) | 0.046 (0.0370)
  22 hours, n=48, 32, 30, 30 | -0.042 (0.0294) | 0.116 (0.0345) | 0.124 (0.0353) | 0.155 (0.0351)
  23 hours, n=48, 32, 30, 30 | -0.042 (0.0310) | 0.168 (0.0365) | 0.137 (0.0374) | 0.157 (0.0371)
  24 hours, n=48, 32, 30, 30 | -0.015 (0.0305) | 0.168 (0.0358) | 0.165 (0.0367) | 0.165 (0.0364)
  25 hours, n=48, 32, 30, 29 | 0.018 (0.0272) | 0.170 (0.0317) | 0.166 (0.0323) | 0.192 (0.0322)

ADVERSE EVENTS:
Time Frame: On-treatment adverse events (AEs), defined as those events occurring while participants were on double-blind treatment, up to and including the day after the last dose in each treatment period (up to 19 weeks), are reported.
Arm/Group | Placebo | FF/VI 50/25 µg | FF/VI 100/25 µg | FF/VI 200/25 µg
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/34 | 0/33 | 0/31
Other Adverse Events (participants affected / at risk) | 2/51 | 4/34 | 4/33 | 3/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=51) | FF/VI 50/25 µg (N=34) | FF/VI 100/25 µg (N=33) | FF/VI 200/25 µg (N=31)
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Caustic injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Raynaud's phenomenon (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.